CLINICAL TRIAL: NCT03565822
Title: Qualitative Study of the Impact of the Birth of a Child With a Rare Abdomino-thoracic Malformation on the Parental Adjustment of the First Year
Brief Title: The Impact of the Birth of a Child With a Rare Abdomino-thoracic Malformation
Acronym: INEMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: University of Lille Nord de France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015_93; 2016-A02050-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-04-24; First posted 2018-06-21 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Congenital Malformation
Keywords: Oesophageal Atresia; Congenital Diaphragmatic Hernia; Short Bowel Syndrome
MeSH Terms: conditions — Congenital Abnormalities; Esophageal Atresia; Hernias, Diaphragmatic, Congenital; Short Bowel Syndrome | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interview (Other): There are two data collection phases (individual interviews +/- focus groups) with parents of children with esophageal atresia, congenital diaphragmatic hernia or short bowel syndrome.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — individual interview and/or focus group Grounded theory qualitative analysis of data related to socio-demographic and child characteristics data First, data will be prepared for qualitative analysis. Digital audio files from the focus groups will be transcribed verbatim and questionnaire data will be entered into an Excel/word data file. Second, focus group data will be qualitatively analyzed using the constant comparative process. A qualitative data analysis program, NVivo11 (Victoria, Australia/ QSR International)) will be used to assist with this coding process.

SUMMARY:
Qualitative study in psychology whose main objective is to propose a grounded theory to report the dynamics of parental adjustment for the period from the announcement of the diagnosis to one year of the child affected by a rare thoracic abdominal congenital malformation, requiring neonatal surgery.

ELIGIBILITY:
Inclusion Criteria:

* to be the parent of a child aged 12 to 36 months old having undergone neonatal surgery following oesophageal Atresia, congenital diaphragmatic hernia or short bowel syndrome diagnosis.
* to have lived with the child during his first year of life
* to have social security coverage
* to speak french

Exclusion Criteria:

* to be a person not having the capacity to consent or enjoying social protection (tutorship or guardianship);
* to be a person deprived of liberty;
* to be a minor;
* to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Level of the dynamics parental adjustment for the period from the announcement of the diagnosis to one year of the child with a rare abdominothoracic malformation requiring neonatal surgery. | at 1 year
  Measure Qualitative Interviews by Grounded theory. The experience with the information received on the disease, describing the socio-demographic characteristics of parents and children with malformation

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Michaud, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, CHU, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided